CLINICAL TRIAL: NCT03719001
Title: A Pilot Study to Evaluate the Effect of Changing Physiological Conditions on the Amplitude and/or Frequency of Myogenic Oscillations
Brief Title: Effect of Changing Physiological Conditions on Myogenic Oscillations: Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PT1802
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases | interventions — Phenylephrine; Dexmedetomidine; clevidipine; Calcium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phenylephrine (Experimental): Phenylephrine (100 ug/ml) infusion will be used to increase blood pressure by 20 mmHg
  Interventions: Drug: Phenylephrine
- Dexmedetomidine (Experimental): Dexmedetomidine infusion will be used to increase blood pressure by 20 mmHg
  Interventions: Drug: Dexmedetomidine
- Clevidipine (Experimental): Clevidipine infusion will be used to increase blood pressure by 20 mmHg
  Interventions: Drug: Clevidipine
- Calcium Chloride (Experimental): Calcium Chloride will be administered to increase blood pressure and to increase blood calcium concentration
  Interventions: Drug: Calcium Chloride
- tetanic stimulus (Experimental): A 5 second 70 mA tetanic stimulus will be used to increase peripheral vascular tone
  Interventions: Other: tetanic stimulus
- Increased venous pressure (Experimental): A 5 minute inflation of a noninvasive blood pressure cuff to 30 mmHg to increase venous pressure in the arm.
  Interventions: Other: Increased venous pressure

INTERVENTIONS:
Drug: Phenylephrine — blood pressure will be increased or decreased by using one of six interventions: phenylephrine (alpha-1 agonist), dexmedetomidine (alpha-2 agonist), clevidipine (Ca channel blocker, CaCl, tetanic stimulus and increase in venous pressure
  Other Names: Neosynephrine
  Arms: Phenylephrine
Drug: Dexmedetomidine — blood pressure will be increased or decreased by using one of six interventions: phenylephrine (alpha-1 agonist), dexmedetomidine (alpha-2 agonist), clevidipine (Ca
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Clevidipine — blood pressure will be increased or decreased by using one of six interventions: phenylephrine (alpha-1 agonist), dexmedetomidine (alpha-2 agonist), clevidipine (Ca
  Other Names: Cleviprex
  Arms: Clevidipine
Other: tetanic stimulus — A 5 second 70 mA tetanic stimulus will be applied to elicit peripheral vasoconstriction (stress response)
  Arms: tetanic stimulus
Other: Increased venous pressure — A 5 minute inflation of a noninvasive blood pressure cuff to 30 mmHg to increase venous pressure in the arm with the pulse oximeter probes.
  Arms: Increased venous pressure
Drug: Calcium Chloride — CaCl will be administered to increase blood pressure and plasma calcium concentration
  Arms: Calcium Chloride

SUMMARY:
Spontaneous myogenic oscillations will be studied under general anesthesia using finger photoplethysmography. This pilot study will explore potential physiological conditions that will effect the amplitude and/or frequency of myogenic oscillations.

DETAILED DESCRIPTION:
This is a single center, nonrandomized, nonblinded, interventional clinical pilot research study that plans to enroll 40 patients.

Study will be conducted while subjects are under general anesthesia.

Myogenic oscillations will be measured using finger photoplethysmography. Changes in the amplitude and/or frequency of these oscillations will be analyzed in response to the interventions. Arterial blood pressure will be recorded to verify the efficacy of the interventions.

Six different interventions that will either lower or increase blood pressure will be applied to the subjects. Each subject will receive 1 or 2 of the six interventions. Each of the 6 interventions will be applied to 8 subject.

The interventions that the subject will not be randomized. They will be determined by the subjects blood pressure immediately before the intervention to guarantee that the blood pressure manipulations are within a safe range.

Data will be analyzed offline using Matlab.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 yrs of age
2. Undergoing surgery in Moffitt-Long operating rooms
3. Receiving general anesthesia
4. Will have an intra-arterial catheter for clinical purposes
5. Able to consent in english

Exclusion Criteria:

1. Under 18 years of age
2. unable to provide informed consent
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
myogenic oscillations | up to 5 minutes
  change in amplitude and/of frequency of myogenic oscillations

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Talke, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No